CLINICAL TRIAL: NCT04404114
Title: Shear Wave Elastography in Differentiating Acute or Chronic Kidney Disease
Acronym: CKD-SWE
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001091RINC
Record Dates: First submitted 2020-04-28; First posted 2020-05-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Elastography; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal renal function: Normal renal function
  Interventions: Diagnostic Test: Shear wave elastography to distinguish AKI from normal kidney
- Acute kidney injury in normal kidney: Acute kidney injury in normal kidney
  Interventions: Diagnostic Test: Shear wave elastography to distinguish AKI from normal kidney
- Acute kidney injury in chronic kidney disease: Acute kidney injury in chronic kidney disease
  Interventions: Diagnostic Test: Shear wave elastography to distinguish AKI from CKD
- Chronic kidney disease: Chronic kidney disease
  Interventions: Diagnostic Test: Shear wave elastography to distinguish CKD from normal kidney

INTERVENTIONS:
Diagnostic Test: Shear wave elastography to distinguish AKI from normal kidney — Record the patient's kidney size, cortical thickness, possible lesion by ordinary renal sonography as well as cortical elasticity by shear wave elastography
  Groups: Acute kidney injury in normal kidney; Normal renal function
Diagnostic Test: Shear wave elastography to distinguish AKI from CKD — Record the patient's kidney size, cortical thickness, possible lesion by ordinary renal sonography as well as cortical elasticity by shear wave elastography
  Groups: Acute kidney injury in chronic kidney disease
Diagnostic Test: Shear wave elastography to distinguish CKD from normal kidney — Record the patient's kidney size, cortical thickness, possible lesion by ordinary renal sonography as well as cortical elasticity by shear wave elastography
  Groups: Chronic kidney disease

SUMMARY:
Chronic kidney disease is a common global public health issue and its prevalence increased year by year. Early diagnosis and intervention can prevent further complications and comorbidities of long-term dialysis, cardiovascular events and mortality as well as improve the patients' life quality. To differentiate acute from chronic kidney disease was crucial especially in the setting of crowded and high-risk emergency department. To diagnose acute or chronic kidney disease, physicians usually use blood sample test combined with image studies such as conventional sonography, CT and MRI. However, there was lots of limited factors. The patients may have no previous visit records, poor renal function to receive contrast medium, or critical clinical condition to undergo time-wasting exam. Although the conventional renal sonography is accessible and inexpensive, the judgement is subjective and provide little clinical information. Recent researches of shear wave elastography in evaluating renal parenchymal stiffness showed some correlation with nephropathy. In our study, aiming to facilitating clinical implication, the investigators will use swear-wave elastography combined with conventional renal sonography to benefit patients in diagnosis of acute or chronic kidney disease.

DETAILED DESCRIPTION:
This is a case-control study. The investigators obtained data from participants who were older than 20 years old and received renal sonography examination in the emergency department of National Taiwan University Hospital. The investigators examined the participants' kidneys by recording the kidney size, cortical thickness, possible lesions and elasticity by shear-wave elastography. These data combined with the participants' medical history and renal function revealed by blood examination will be analyzed. This study was designed to determine the correlation between renal cortical elasticity and chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* The patients older than 20 years old who needed to receive renal sonography in emergency department of National Taiwan University Hospital.

Exclusion Criteria:

* The patients who didn't obtain agreement.
* The patients who can't cooperate or follow the directions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 400 patients with normal kidney function and 400 patients with abnormal kidney function
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the correlation of kPa ratio and renal function in chronic renal disease | change in renal function after 2 weeks
  The analysis will be conducted to determine the correlation between kPa ratio measured by elastography and renal function in patients with chronic renal disease

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan